CLINICAL TRIAL: NCT07246044
Title: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) Targeting the Primary Somatosensory Cortex for Bipolar Depression in Adolescents: A Randomized Double-Blind Controlled Trial
Brief Title: HD-tDCS for Adolescent Bipolar Depression Targeting S1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Principal Investigator, Fei Wang, Professor, Jiangsu Province Nanjing Brain Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81725005-10
Record Dates: First submitted 2025-09-18; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adolescent; Bipolar Depression; tDCS; Primary Somatosensory Cortex; Bipolar Disorder Depression
Keywords: primary somatosensory cortex; adolescent; bipolar depression; high-definition transcranial direct current stimulation
MeSH Terms: conditions — Bipolar Disorder | interventions — Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HD-tDCS Targeting Right S1 (Experimental): Participants in this arm will receive active HD-tDCS targeting the right S1. Anodal stimulation will be delivered at the C4 position according to the international 10-20 EEG system, with cathodes placed at FC4, C6, C2, and CP4. The current intensity is set at 2.0 mA for 20 minutes per session, administered twice daily for 10 days (total of 20 sessions). Participants received stable pharmacological treatment during the intervention period.
  Interventions: Device: Active HD-tDCS; Drug: Antipsychotics, mood stabilizers, etc.
- Sham Stimulation at Right S1 (Sham Comparator): Participants in this arm will receive sham HD-tDCS using the same electrode configuration as the active group (anode at C4; cathodes at FC4, C6, C2, and CP4), but without delivering effective current after the initial ramp-up. The sham stimulation mimics the sensation of real stimulation without physiological effects. Sessions will be delivered twice daily for 10 days (total of 20 sessions). Participants received stable pharmacological treatment during the intervention period.
  Interventions: Drug: Antipsychotics, mood stabilizers, etc.; Device: Sham HD-tDCS

INTERVENTIONS:
Device: Active HD-tDCS — HD-tDCS is a non-invasive neuromodulation therapy which has been recognized as a helpful treatment for depression. During each HD-tDCS treatment, the electrode field is generated by a 4*1 ring montage which is placed over the scalp on the brain region of interest with an electrical current induced to modulate brain activity.
  Arms: Active HD-tDCS Targeting Right S1
Drug: Antipsychotics, mood stabilizers, etc. — During the HD-tDCS treatment period, all the participants will maintain the stable medication regimen according to clinical practice guidelines.
Device: Sham HD-tDCS — Sham HD-tDCS is administered using the same electrode configuration as the active HD-tDCS condition. During each session, the device ramps up current briefly (typically 30 seconds) to mimic the initial sensation of stimulation, then remains off for the remainder of the 20-minute session. This method produces the same tactile perception as active stimulation without delivering a therapeutic dose of current.
  Arms: Sham Stimulation at Right S1

SUMMARY:
This randomized, double-blind, sham-controlled clinical trial aims to evaluate the efficacy and underlying biological mechanisms of HD-tDCS targeting the primary somatosensory cortex in adolescents with bipolar depression. Participants will be randomly assigned to receive either active HD-tDCS or sham stimulation, in addition to routine clinical care. Biological data, including neuroimaging, blood biomarkers, voice and facial features, Photoplethysmography (PPG), Electroencephalography (EEG), and behavioral data, will be collected to explore potential predictors of treatment response.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and underlying biological mechanisms of HD-tDCS targeting the primary somatosensory cortex (S1) in adolescents with bipolar depression. Participants will be randomly assigned (1:1) to receive either active HD-tDCS or sham stimulation for 10 consecutive days (twice daily, 20 minutes each session), in addition to standard clinical care.

Multimodal assessments will be conducted at baseline, mid-treatment (after 10 sessions), and post-treatment, including clinical symptom scales, neurocognitive evaluations, structural and functional MRI, blood biomarkers (15ml of peripheral blood), as well as digital phenotyping data such as voice, EEG, PPG, sleep, and behavioral metrics.

The study also aims to identify objective biomarkers predictive of treatment response and to elucidate the neurobiological mechanisms associated with HD-tDCS applied to the S1 region. All procedures including MRI, tDCS, and assessments are non-invasive and free of charge for participants. The total duration of data collection and follow-up is expected to span approximately two years.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 18 years of age;
* Participants fulfill the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria for bipolar disorder (BD). Participants are assessed by the Structured Clinical Interview for DSM-IV for Axis I Disorders (SCID-I, patients' age ≥18 years old), or the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (K- SADS-PL, patients' age< 18 years old);
* A current moderate or severe depressive episode defined by HAMD≥17 and Young Mania Rating Scale (YMRS) <12;
* Participants receive a stable psychotropic medication regimen prior to randomization to the trial and are willing to remain on the stable regimen during the HD-tDCS treatment phase;
* Participants and 1 or 2 parents (patients' age< 18 years old) provide informed consent after the detailed description of the study.

Exclusion Criteria:

* Prior rTMS or tDCS or electroconvulsive therapy (ECT) treatment or standard psychological therapy within 6 months prior to screening;
* Comorbidity of other DSM-IV axis I disorders or personality disorders;
* Judged clinically to be at serious suicidal risk;
* Diabetes mellitus, hypertension, vascular and infectious diseases and other major medical comorbidities;
* Unstable medical conditions, e.g., severe asthma;
* Neurological disorders, e.g., history of head injury with loss of consciousness for ≥ five minutes, cerebrovascular diseases, brain tumors and neurodegenerative diseases;
* Mental retardation or autism spectrum disorder;
* Contraindications to MRI (e.g., severe claustrophobia, pacemakers, metal implants);
* Contraindications to tDCS (e.g., metal in head, history of seizure, EEG test suggesting high risk of seizure, known brain lesion);
* Current drug/alcohol abuse or dependence;
* Pregnant or lactating female.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by the 17-item Hamilton Depression Rating Scale (HAMD-17) at Week 2. | Baseline and after 2 weeks.
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 17 or higher indicate moderate, severe, or very severe depression.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms assessed by HAMD-17 after week 1. | Baseline and after 1 week.
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 17 or higher indicate moderate, severe, or very severe depression.
Change in anxiety symptoms assessed by Hamilton Anxiety Rating Scale (HAMA) after week 1 and after week 2. | Baseline, after 1week and after 2 weeks.
  The HAMA consists of 14 items designed to assess the severity of a patient's anxiety. Each item is rated on a scale of 0 (not present) to 4 (severe), with a total score ranging from 0 to 56. Higher scores indicate greater anxiety. Change in total score from baseline will be calculated.
Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) after week 1 and after week 2. | Baseline and after 1 week and after 2 weeks.
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) after 1 week and after 2 week. | Baseline, after 1 week and after 2 weeks.
  MADRS is a clinician-rated scale used to assess depressive symptom severity and detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is rated from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). The total score of MADRS ranges from 0 to 60, with higher score indicating more severe depression.
Change in brain functional connectivity measured by resting-state functional MRI | Baseline, after 1 week and after 2 weeks.
  Resting-state functional magnetic resonance imaging (rs-fMRI) will be used to assess changes in the connectivity of the primary S1 and associated networks.
Change in Cytokines (reported in pg/mL) | Baseline, after 1 week, and after 2 weeks.
  Peripheral blood biomarkers will be measured to evaluate inflammatory and immune responses to HD-tDCS treatment.
  Interferon-α (IFN-α) Interferon-γ (IFN-γ) Interleukin-1β (IL-1β) Interleukin-2 (IL-2) Interleukin-4 (IL-4) Interleukin-5 (IL-5) Interleukin-6 (IL-6) Interleukin-8 (IL-8) Interleukin-10 (IL-10) Interleukin-17 (IL-17) Tumor necrosis factor-alpha (TNF-α)
Change in Immune-inflammatory ratios (unitless) | Baseline, after 1 week, and after 2 weeks.
  Platelet-to-lymphocyte ratio (PLR) Neutrophil-to-lymphocyte ratio (NLR) Monocyte-to-HDL cholesterol ratio (MHR) These biomarkers are selected to reflect systemic inflammatory activity and immune status.
Adverse events and tolerability of HD-tDCS | Baseline, after 1 week and after 2 weeks
  Adverse events related to HD-tDCS will be monitored throughout the treatment period. Participants will be evaluated for scalp irritation, headache, dizziness, fatigue, or other discomforts after each session. Severity and frequency will be recorded using a standardized adverse event form.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Study Chair — the Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No